CLINICAL TRIAL: NCT06939205
Title: The Impact of Different Body Surface Area Prediction Equations on Ventricular Dilatation Prevalence in Youth Soccer Players
Brief Title: Body Surface Area Prediction Impacts on Ventricular Dilatation Prevalence
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Alessandro Minetto, Full Professor, University of Turin, Italy
Other Study IDs: UniTO&JMedBSAstudy
Record Dates: First submitted 2025-04-03; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiomyopathies
Keywords: 3-D optical imaging; Body surface area; soccer; transthoracic echocardiography
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Assessment of body surface area and assessment ventricular dilatation prevalence — Estimation of body surface area and quantification of absolute and relative values of echocardiographic variables

SUMMARY:
The goals of this observational study are to investigate the accuracy of different predictive equations for body surface area (BSA) estimation and to evaluate the impact of different BSA normalizations on ventricular dilatation prevalence in youth soccer players. Two convenience samples of young soccer players of both genders will be recruited. Acquisition of optical images (for the players of the first sample), two-dimensional echocardiographic assessment (for the players of the second sample), and weight and height measurements (for the players of both samples) will be performed. BSA estimates will be derived from optical images (for the players of the first sample) and from ten different predictive equations obtained from the literature (for the players of both samples). Comparisons between optical imaging - derived BSA and BSA estimates obtained with the ten predictive equations will be performed for the players of the first sample. Absolute and relative values of different echocardiographic variables will be considered for the players of the second sample to assess the ventricular dilatation prevalence.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* regular sports participation

Exclusion Criteria:

- athletic heart syndrome

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Soccer players of both genders
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Body surface area (BSA) | Baseline (preseason investigation)
  Estimation of the BSA value: weight (unit of measurement: kg) and height (unit of measurement: m) will be combined to report BSA in m^2
Left ventricular dilatation prevalence | Baseline (preseason investigation)
  Absolute and relative (normalized to body surface area - BSA) values of the following echocardiographic variables will be considered:
  1) left ventricular end-diastolic diameter (LVEDD: absolute value in mm; relative value in mm/m^2); 2) left ventricular end diastolic volume (LVEDV: absolute value in ml; relative value in ml/m^2).
  The left ventricular dilatation will be identified if one or both the relative variables are above the following cut-points: i) LVEDD: 30 mm/m^2 for males and 31 mm/m^2 for females; ii) LVEDV: 74 ml/m^2 for males and 61 ml/m^2 for females.
Right ventricular dilatation prevalence | Baseline (preseason investigation)
  Absolute and relative (normalized to body surface area - BSA) values of the fright ventricular basal diameter (RVBD: absolute value in mm; relative value in mm/m^2) will be considered.
  The right ventricular dilatation will be identified if RVBD is above the cut-point of 22 mm/m^2 for both males and females

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alessandro Minetto, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin, Torino, Italy

IPD SHARING:
Plan to Share IPD: No